CLINICAL TRIAL: NCT05672030
Title: Role of Interleukin 5 (IL-5) and IL-5R Signaling in Non-eosinophil Upper Airway Cells in Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Role of IL-5R Signaling in Non-eosinophil Upper Airway Cells in CRSwNP
Acronym: RECAP-5
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tanya Laidlaw, MD, Associate Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2003P002088
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nasal Polyps; Aspirin-exacerbated Respiratory Disease
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aspirin-exacerbated respiratory disease (AERD): Aspirin-exacerbated respiratory disease (AERD)
  Interventions: Other: Non-Interventional
- Aspirin-tolerant chronic rhinosinusitis with nasal polyps (CRSwNP): Aspirin-tolerant chronic rhinosinusitis with nasal polyps (CRSwNP)
  Interventions: Other: Non-Interventional
- Healthy controls: Individuals who do not have AERD or CRSwNP
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — No intervention.

SUMMARY:
The overarching hypothesis of this proposal is that IL-5 acts on multiple sinus tissue cell types, including plasma cells and epithelial cells, to promote immune dysregulation, and that inhibition of IL-5 affects several relevant effector pathways that lead to clinical benefit.

DETAILED DESCRIPTION:
Further characterization of the role of IL-5Rα expression and function on human plasma cells will determine whether inhibiting IL-5 signaling on these cells offers therapeutic promise in other diseases related to plasma cell proliferation. Further characterization of human upper airway epithelial cell IL-5Rα expression and function will determine whether or not inhibiting IL-5 signaling on these cells offers therapeutic promise in other diseases related to epithelial dysfunction. IL-5Rα expression has been identified on several relevant sinus tissue effector cells, including on nasal polyp plasma cells and epithelial cells, and the aim of this study is to further the field by determining the consequences of IL-5 signaling on those cells.

ELIGIBILITY:
Inclusion Criteria:

* AERD, CRSwNP, healthy controls

Exclusion Criteria:

* Not on any systemic steroids or respiratory biologics at time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AERD, CRSwNP, healthy controls undergoing planned elective sinus surgery.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Laidlaw, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Full Range); unit: years] | 54 [25 to 69] | 52 [27 to 64] | 49 [23 to 66] | 52 [23 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 7 | 18
  Male | 4 | 5 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 8 | 8 | 7 | 23
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Nasal Polyp Plasma Cell Transcriptome
Description: We will determine the number of participants from whom a transcriptional profile of nasal polyp plasma cells is analyzable from bulk RNA sequencing of sorted nasal polyp plasma cells.
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

2. Secondary Outcome: Number of Participants With Functional Readouts of IL-5Ra on Nasal Polyp Plasma Cells.
Description: We will determine the number of participants from whom a readout of IL-5Ra is analyzable from the plasma cells in their nasal tissue
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

3. Secondary Outcome: Number of Patients for Whom IL-5Ra Signaling on Nasal Epithelial Cells Can be Analyzed
Description: We will determine the number of participants from whom IL-5-elicited signaling on their nasal epithelial tissue can be analyzed.
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls
Number analyzed (Participants) | 10 | 10 | 10
Participants | 10 | 10 | 10

ADVERSE EVENTS:
Time Frame: At the single visit at which samples were collected. This was a single-visit sample-collection observational study. No intervention.
Arm/Group | Aspirin-exacerbated Respiratory Disease (AERD) | Aspirin-tolerant Chronic Rhinosinusitis With Nasal Polyps (CRSwNP) | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT05672030/Prot_SAP_000.pdf